CLINICAL TRIAL: NCT02936258
Title: A Phase III Multi-centre Open-label Randomized Controlled Trial of Multi-parametric Magnetic Resonance Imaging (MRI)-Targeted Biopsy Compared to Systematic Trans-rectal Ultrasound (TRUS) Guided Biopsy
Brief Title: PRostate Evaluation for Clinically Important Disease: MRI vs Standard Evaluation Procedures
Acronym: PRECISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: Ontario Institute for Cancer Research (Other); Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRECISE Trial
Record Dates: First submitted 2016-09-28; First posted 2016-10-18 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI (Other): Men in Arm A will undergo a MRI followed by either a targeted biopsy of suspicious areas or will be followed for two years if there is no suspicious areas identified by MRI. The unbiopsied men will have a repeat MRI at 2 years.
  Interventions: Procedure: MRI; Procedure: MRI Targeted Biopsy
- Standard of Care (Active Comparator): Men in Arm B will undergo a 12-core systematic TRUS guided biopsy. All men in the study will be followed for two years or until they have had radical treatment (whichever comes first).
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Standard of Care — Men in Arm B will undergo a 12-core systematic TRUS guided biopsy. All men in the study will be followed for two years or until they have had radical treatment (whichever comes first).
  Arms: Standard of Care
Procedure: MRI — Men will undergo a MRI followed by either a targeted biopsy of suspicious areas or will be followed for two years if there is no suspicious areas identified by MRI.
  Arms: MRI
Procedure: MRI Targeted Biopsy — Men will undergo a MRI followed by either a targeted biopsy of suspicious areas or will be followed for two years if there is no suspicious areas identified by MRI.
  Arms: MRI

SUMMARY:
The aim of this study is to assess the efficacy of MRI-targeted biopsy compared to standard of care systematic TRUS guided biopsy in the detection of clinically significant and clinically insignificant prostate cancer in men without prior biopsy. The implication of this trial is that MRI-targeted biopsy could replace systematic TRUS guided biopsy as the standard of care in the diagnosis of prostate cancer.

DETAILED DESCRIPTION:
The standard pathway for prostate cancer diagnosis is trans-rectal ultrasound guided (TRUS) biopsy of the prostate following an elevated PSA. TRUS guidance is performed primarily for anatomic guidance as the ultrasound poorly discriminates between cancerous and non-cancerous tissue. TRUS guided prostate biopsies are concentrated in areas of the peripheral zone, thought to harbor the majority of cancer.

An alternative pathway for prostate cancer diagnosis in men with elevated PSA is to perform multi-parametric magnetic resonance imaging (MPMRI) to localize cancer. This information is used to direct a subsequent biopsy, known as an MRI-targeted biopsy. MRI-targeted biopsy has been shown in preliminary studies to detect a similar or greater amount of clinically significant cancer than systematic TRUS guided biopsy and has several other potential advantages including: the ability to differentiate between clinically significant and insignificant cancer, reducing unnecessary biopsy and fewer numbers of biopsy cores, reducing biopsy-related side-effects.

A 'clinically insignificant cancer' is cancer that is unlikely to progress or to affect an individual's life expectancy and therefore does not warrant treatment. However when diagnosed with low grade cancer that is likely to be insignificant, a large proportion of subjects request treatment in case a more significant cancer is present. A challenge in this area is that subjects are typically not aware that their cancer is clinically insignificant, and often view the early diagnosis and aggressive treatment they have been subjected to as life-saving.

A prostate cancer detection procedure that differentiates clinically significant cancer from clinically insignificant cancer is therefore a major unmet need.

The potential implications of this trial include:

* A redefinition of the prostate cancer diagnostic pathway;
* A reduction in the number of subjects undergoing prostate biopsy;
* A reduction in the number of biopsy cores taken per subject;
* A reduction in biopsy-related adverse events including sepsis and pain;
* A reduction in the over-diagnosis of clinically insignificant prostate cancer;
* A reduction in the economic burden of diagnosing and treating prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible, all inclusion criteria must be met:

1. Men at least 18 years of age referred with clinical suspicion of prostate cancer who have been advised to have a prostate biopsy;
2. ≥5% chance of high-grade prostate cancer as calculated using individualized risk assessment of prostate cancer calculator, PCPTRC 2.0, found at http://deb.uthscsa.edu/URORiskCalc/Pages/calcs.jsp;
3. Serum PSA ≤ 20ng/ml within 3 months of randomization
4. Fit to undergo all procedures listed in protocol;
5. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy
2. Prior treatment for prostate cancer
3. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated GFR ≤ 50mls/min)
4. Contraindication to prostate biopsy
5. Men in whom artifact would reduce the quality of the MRI, i.e. previous hip replacement surgery, metallic hip replacement or extensive pelvic orthopaedic metal work
6. Unfit to undergo any procedures listed in protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
MRI-The proportion of men with clinically significant cancer (Gleason > 7) | 1 year
  To determine whether the proportion of men with clinically significant cancer (Gleason > 7) detected by MRI-targeted biopsy is no less than systematic TRUS guided biopsy.

SECONDARY OUTCOMES:
Biopsy-The proportion of men with clinically significant cancer (Gleason ≥7) | 1 year
  1. The proportion of men with clinically significant cancer (Gleason ≥7) detected by MRI-targeted biopsy is greater than systematic TRUS guided biopsy.
Proportion of men in each arm with clinically insignificant cancer | 1 year
Proportion of men in each arm with Gleason >4+3 detected. | 1 year
Proportion of men in MRI arm who avoid biopsy. | 1 year
Proportion of men in the MRI arm whom the PI-RADS score for suspicion of clinically significant cancer was 3, 4 or 5 but no clinically significant cancer was detected. | 1 year
Proportion of men in each arm who go on to definitive local treatment (e.g. radical prostatectomy, radiotherapy, brachytherapy) or systemic treatment (e.g. hormone therapy, chemotherapy). | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - London Health Sciences Centre-Victoria Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS du Centre-Ouest-de-I'ile-de-Montreal-Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Plan to share publication

REFERENCES:
- [Derived] Klotz L, Chin J, Black PC, Finelli A, Anidjar M, Machado A, Levental M, Ghai S, Chang SD, Patel C, Kassam Z, Loblaw A, Kebabdjian M, Pond G, Haider MA. Magnetic Resonance Imaging-Targeted Versus Systematic Prostate Biopsies: 2-year Follow-up of a Prospective Randomized Trial (PRECISE). Eur Urol Oncol. 2024 Jun;7(3):456-461. doi: 10.1016/j.euo.2023.09.013. Epub 2023 Oct 12. PMID 37838556
- [Derived] Klotz L, Chin J, Black PC, Finelli A, Anidjar M, Bladou F, Mercado A, Levental M, Ghai S, Chang SD, Milot L, Patel C, Kassam Z, Moore C, Kasivisvanathan V, Loblaw A, Kebabdjian M, Earle CC, Pond GR, Haider MA. Comparison of Multiparametric Magnetic Resonance Imaging-Targeted Biopsy With Systematic Transrectal Ultrasonography Biopsy for Biopsy-Naive Men at Risk for Prostate Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):534-542. doi: 10.1001/jamaoncol.2020.7589. PMID 33538782